CLINICAL TRIAL: NCT00437229
Title: An Open-Label, Phase I Study to Assess the Pharmacokinetic Interaction Between Repeat Doses of Oral Casopitant and Intravenous and Oral Doses of Dexamethasone and Intravenous and Oral Doses of Ondansetron When Administered in Healthy Adult Subjects
Brief Title: A Study to Assess the Safety & Interaction Between GW679769, Dexamethasone, & Ondansetron When Taken by Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NKV100787
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Nausea and Vomiting, Chemotherapy-Induced
Keywords: GW679769,; Casopitant,; Dexamethasone,; Healthy Human Volunteer; Ondansetron,
MeSH Terms: conditions — Nausea; Vomiting | interventions — casopitant; Dexamethasone; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects in Part A (Experimental): In PART A, subjects received Regimen A: oral casopitant alone (150 mg once daily [QD] Day 1, 50 mg QD Days 2 and 3); Regimen B: oral dexamethasone (20 mg QD Day 1 and 8 mg twice daily [BID] Days 2 and 3) and intravenous (IV) ondansetron (32 mg single-dose Day 1); and Regimen C: oral casopitant as in Regimen A, IV ondansetron as in Regimen B and a lower dose oral dexamethasone than in Regimen B (12 mg QD Day 1, 8 mg QD Days 2 and 3).
  Interventions: Drug: Casopitant (GW679769) Oral Tablets; Drug: dexamethasone; Drug: ondansetron
- Subjects in Part B (Experimental): In PART B, subjects received Regimen D: oral casopitant alone (150 mg QD Day 1, 50 mg QD Days 2 and 3); Regimen E: IV dexamethasone (8 mg single-dose Day 1 only) and oral ondansetron (8 mg BID Days 1 to 3); and Regimen F: oral casopitant regimen as in Regimen D, and IV dexamethasone and oral ondansetron as in Regimen E.
  Interventions: Drug: Casopitant (GW679769) Oral Tablets; Drug: dexamethasone; Drug: ondansetron

INTERVENTIONS:
Drug: Casopitant (GW679769) Oral Tablets — Casopitant (GW679769) tablets will be available as white, film-coated tablets containing 50 mg of GW679769 as the mesylate salt for oral administration.
Drug: dexamethasone — Dexamethasone will be available as 4 mg tablets for oral administration and injection for IV administration.
Drug: ondansetron — Ondansetron for oral use will be available as 8 mg tablets to be taken with 240 milliliters (mL) of water on an empty stomach. For IV use, ondansetron 32 mg will be infused intravenously over a period of 15 minutes.
  Other Names: GW679769 Oral Tablets; dexamethasone oral tablets & intravenous; ondansetron oral tablets & intravenous

SUMMARY:
GW679769 may affect liver enzymes that metabolize dexamethasone and ondansetron. This study is designed to test the safety and the extent of the GW679769 affect on dexamethasone and ondansetron levels in humans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males or females
* Age: 18 to 55 years, inclusive
* A female subject who is non-childbearing potential or using acceptable contraceptive methods.
* Adequate organ systems function
* Able to swallow and retain oral medication
* Able to understand and comply with protocol requirements and instruction and is likely to complete the study.

Exclusion Criteria:

* Cannot participation if subject has a clinically relevant abnormality, medical condition, or circumstance that makes them unsuitable for the study per the study doctor.
* History of drug or other allergy which, in the opinion of the Investigator, contraindicates participation.
* Use of an investigation drug within 28 days or 5 half-lives.
* Blood donation in excess of 500mL within 56 days prior to dosing or intends to donate within 30 days of the post-treatment follow-up visit.
* Presence of or suspected iron deficiency
* Positive stool for occult blood
* Female subject who is lactating
* Positive urine drug screen
* Positive for HIV antibody, hepatitis C antibody or hepatitis B surface antigen
* Use of tobacco-containing products within the past 12 months prior to screening
* History of drug or alcohol abuse or dependence within 6 months of screening
* History or presence of uncontrolled emesis
* Positive purified protein derivative (PPD) skin test for tuberculosis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2007-02-19 (Actual); Primary Completion 2007-05-15 (Actual); Study Completion 2007-05-15 (Actual)

PRIMARY OUTCOMES:
Part A: Period 1 & 2: Plasma levels of casopitant, dexamethasone, & ondansetron will be checked on Day 1, 2 and/or 3. Part B: Period 1, 2 & 3: Plasma levels of casopitant, dexamethasone, & ondansetron will be checked on Day 1, 2 and/or 3. | checked on Day 1, 2 and/or 3

SECONDARY OUTCOMES:
Safety is evaluated by: Clinical Lab Tests done | at Screening, Day -1 & Followup.
Vitals Signs taken & Adverse Events monitored | at each visit starting at Day -1.
12 lead ECGs & Serum Pepsinogen level tests | at Screening & Followup.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

REFERENCES:
- [Background] Johnson B, Adams L, Lu E, Zhang K, Lebowitz P, Lates C, Blum R. Impact of casopitant, a novel NK-1 antagonist, on the pharmacokinetics of ondansetron and dexamethasone. Support Care Cancer. 2009 Sep;17(9):1177-85. doi: 10.1007/s00520-008-0571-5. Epub 2009 Feb 10. PMID 19205755
- See also: Results for study 100787 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/NKV100787?search=study&search_terms=100787#rs